CLINICAL TRIAL: NCT03790384
Title: The Effects of Sequential Mitomycin and Bacillus Calmette-Guérin Treatment Versus Bacillus Calmette-Guérin Monotherapy in Patients With High Risk Non-Muscle Invasive Bladder Cancer
Brief Title: Sequential Combination Therapy in Bladder Cancer
Acronym: MITOBCG
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera "Sant'Andrea" (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-004540-37
Record Dates: First submitted 2018-12-11; First posted 2018-12-31 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Mitomycin; BCG Vaccine

STUDY DESIGN:
Intervention Model Description: The subjects will be assessed for eligibility at the screening visit (Visit 1) three weeks after TURB and re-TURB prior to randomization and only subjects who fulfil the inclusion criteria will be included: patients with a diagnosis of High risk NMIBC: T1 tumor, G3, CIS, or multiple and recurrent and large (>3 cm) Ta or patients in the last EAU recurrence category (EAU/EORTC recurrence score >/=10). Patients selected for the study, are centrally randomized (randomization is performed at the Sant'Andrea Hospital) to receive BCG induction treatment according to the standard protocol (an instillation once a week for six weeks) with ImmuCyst (81 mg Connaught strain BCG). Patients in group two received BCG treatment with the same protocol with a 40 mg mitomycin instillation the day before .
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bacillus Calmette-Guérin (No Intervention): Patients receive Bacillus Calmette-Guérin induction treatment according to the standard protocol (an instillation once a week for six weeks) with ImmuCyst (81 mg Connaught strain BCG).
- Mytomicin and Bacillus Calmette-Guérin (Experimental): Patients received BCG treatment with the same protocol. Intervention will be a 40 mg mitomycin instillation the day before every single BCG instillation
  Interventions: Drug: Mitomycin

INTERVENTIONS:
Drug: Mitomycin — Patients receive BCG induction treatment according to the standard protocol (an instillation once a week for six weeks) with ImmuCyst (81 mg Connaught strain BCG) with a 40 mg mitomycin instillation the day before .
  Other Names: Bacillus Calmette-Guerin
  Arms: Mytomicin and Bacillus Calmette-Guérin

SUMMARY:
A consecutive series of patients with High Risk Non-Muscle Invasive Bladder Cancer will be enrolled in several centres. The subjects will be assessed for eligibility at the screening visit (Visit 1) three weeks after Trans-Urethral Resection of the Bladder (TURB) and re-TURB prior to randomization and only subjects who fulfil the inclusion criteria will be included. Patients selected for the study, are centrally randomized (randomization is performed at the Sant'Andrea Hospital) to receive BCG induction treatment according to the standard protocol (an instillation once a week for six weeks) with Immucyst (81 mg Connaught strain BCG). Patients in group two received BCG treatment with the same protocol with a 40 mg mitomycin instillation the day before .

DETAILED DESCRIPTION:
Methods:

A consecutive series of patients with High Risk Non-Muscle Invasive Bladder Cancer will be enrolled in several centres

Clinical evaluation:

Patients with High Risk Non-Muscle Invasive Bladder Cancer will be enrolled. For each patients we evaluate the following parameters:

* Age
* Sex
* Occupational status
* Smoker Status
* Co-morbidities
* Concomitant medications or treatment
* Height, Weight, BMI
* Urinary symptoms evaluation:

  * Presence of Haematuria at the diagnosis
  * International Prostatic Symptoms Score
* Laboratories Analyses

  * Hemoglobin serum level
  * Creatinine
* EORTC/EAU risk stratification
* Endoscopic bladder evaluation (video-recorded and centrally evaluated)

  * Number of Tumors
  * Diameter of Tumors (<3 cm or > 3 cm)
  * Location of Bladder Tumors
* TURB (video recorded) + histological examination
* Re-TURB showing no evidence of neoplasms
* Follow-up

  * Cystoscopy (video will be recorded and centrally re-evaluated for recurrence) and cytology every three months later
  * Recurrence Rate
  * Number of Recurrence Rate
  * Number of Tumors
  * Diameter of Tumors
  * Location of Bladder Tumors
  * Urethral Stricture
  * Bladder mapping at 6 months
  * Uro Tomography Computerized yearly

Intervention:

The subjects will be assessed for eligibility at the screening visit (Visit 1) three weeks after TURB and re-TURB prior to randomization and only subjects who fulfil the inclusion criteria will be included: patients with a diagnosis of High risk Non Muscle Invasive Bladder Cancer (NMIBC): T1 tumor, G3, Carcinoma in Situ (CIS), or multiple and recurrent and large (>3 cm) Ta or patients in the last EAU recurrence category (EAU/EORTC recurrence score >/=10). Patients selected for the study, are centrally randomized (randomization is performed at the Sant'Andrea Hospital) to receive BCG induction treatment according to the standard protocol (an instillation once a week for six weeks) with Immucyst (81 mg Connaught strain BCG). Patients in group two received BCG treatment with the same protocol with a 40 mg mitomycin instillation the day before .

Adverse Events All the adverse events that will occur in the study will be recorded in the case report form (CRF).

An adverse event (AE) is defined as a harmful clinical event occurring in a patient or a human volunteer involved in a clinical experimentation who received a drug that does not necessarily have a relationship with the treatment given. It is considered AE any medical occurrence including undesirable signs or symptoms or abnormal lab finding.

A Serious Adverse Event (SAE) is an AE that, independently from the dosage of the drug used, had one of the following characteristic:

1. Results in death
2. It's life threatening (i.e. the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe)
3. It's cause of hospital admission or increase the time of hospitalization
4. It's cause of congenital abnormalities at birth
5. It's cause of disability or severe and long lasting inability Treatment Emergent Adverse Events (TEAE) is defined as any event not present prior to the initiation of the treatments or any event already present that worsens in the either intensity or frequency following exposure to the treatments.

A Suspected Unexpected Serious Adverse Reaction (SUSAR) is the term used to refer to an adverse event that occurs in a clinical trial subject, which is assessed as being unexpected, serious and as having a reasonable possibility of a causal relationship with the study drug. It is defined as an untoward and unintended response to a study drug, at any dose, which is not listed in the product information, and meets one of the above mentioned serious characteristics.

Generally AEs are collected after signing the informed consent form and could be related or unrelated to the study drug.

For any AE/SAE recorded during the study a causal relationship with the drug used will be assessed as follows:

* Very likely: the AE/SAE is temporally associated to the drug administration, cannot be explained by other clinical conditions and/or concomitant treatments, disappears with drug withdrawal and recurs after drug reintroduction;
* Likely: the AE/SAE is temporally associated to the drug administration, cannot be explained by other clinical conditions and/or concomitant treatments, disappears with the drug withdrawal. There is no information on drug reintroduction;
* Possible: the AE/SAE is temporally associated to the drug administration, cannot be explained by other clinical conditions and/or concomitant treatments, disappears with drug. There is no information available on the drug withdrawal and reintroduction;
* Doubtful: the AE/SAE could be temporally associated to the drug administration, but can be explained by other clinical conditions and/or concomitant treatments;
* Not correlated: the AE/SAE is not temporally associated to the drug administration and/or can be explained by other clinical conditions and/or concomitant treatments.
* An AE/SAE with causal relationship very likely, likely possible with the drug is considered correlated with it and is defined Adverse Reaction (ADR).

World Health Organization (WHO) defines ADR as "a response to a drug which is noxious & unintended and which occurs at doses normally used for prophylaxis diagnosis or therapy of a disease or for modification of a physiological function".

The difference between AE and ADR is that AE event does not imply causality but not for ADR, a causal rule is suspected.

An ADR unexpected is defined an ADR that for nature and severity is not listed in the product information (Reference Safety Information (RSI)/Investigator's Brochure (IB)).

Toxicity evaluation Urine culture is performed 3 days before each bladder instillation to check urine sterility (mandatory before the first course, optional before the following instillations). Treatment related adverse events are recorded by the patients on a diary.

Outcome analysis: adverse events are self-recorded by the patients after each instillation and classified by the investigator according to a classification grid considering account duration and intensity as proposed by Saint et al. Thus, toxicity is classified as systemic or local and class I (mild) up to class III (severe). The baseline symptoms are also assessed. Local toxicity included bacterial cystitis, BCG induced cystitis, frequency, macroscopic hematuria and "other". Bacterial cystitis is defined as the occurrence of culture proven (not BCG) bacterial cystitis. Irritative bladder symptoms with negative urine culture are classified as BCG induced (chemical) cystitis. "Other" local side effects include granulomatous prostatitis, epididymitis, ureteral obstruction and contracted bladder. Systemic side effects are classified as fever (≥39 °C), influenza like symptoms including general malaise and chills, BCG induced lung infection, liver toxicity, and BCG sepsis. Skin rash, arthralgia and arthritis are classified as possible allergic reactions. Based on the severity of adverse events experienced by the patient, one of the investigator, who is blind to the given therapy, decides whether the next instillation is to be done, postponed, deleted or whether the patient should receive specific anti-tuberculosis therapy. Dose reduction is not allowed in either group. Patients will also complete flow-volume charts for three days after BCG instillations and two questionaries to assess urinary symptoms and patient's perception of bladder pain as the chronic prostatitis symptoms index (NIH-CPSI) and the pelvic pain and urgency/frequency questionaire (PUF). The efficacy of both treatments is assessed at 3, 6,9,12 months with flexible cystoscopy, urinary cytology and bladder biopsy if needed.

STATISTYCAL ANALYSIS Using type I error, and a power of 2.5% and 81% respectively, and by proposing the hypothesis that Immucyst induced a recurrence in about 60% of cases (EORTC risk score 10) and its combination with mitomycin decreases this percent by 30%, it was calculated that 66 subjects per group were necessary to detect this difference using the adjusted chi-square method and Statistical Solution calculator. Student's T test was used for continuous variables. Two-sided p values were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high risk non muscle invasive bladder cancer
* High risk of progression (EORTC risk score > 6)
* Males
* Signature of Informed Consent
* Ability of consent

Exclusion Criteria:

* Low Risk Non-Muscle Invasive Bladder Cancer
* Muscle Invasive Bladder Cancer
* Concomitant Urothelial Bladder Cancer in the Upper-Urinary Tract
* Previous bladder or prostate surgery
* Prostate or bladder radiotherapy
* Urinary tract infection
* Chronic urinary retention or indwelling catheters
* Neurological patients
* Previous BCG infections
* Previous or current chemotherapy for other kind of cancers
* Patients older than 75
* WHO performance status 3-4
* Residual tumour on re-TURB

Min Age: 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-01-15 (Estimated); Primary Completion 2019-09-15 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 2 years
  To evaluate the effect in term of recurrence rate of sequential combination therapy of Mitomycin and Bacillus Calmette-Guérin versus Bacillus Calmette-Guérin monotherapy in patients with High grade Non-Muscle Invasive Bladder Cancer.through cystoscopy every three months and Uro Tomography Computerized yearly

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years
  To evaluate the overall toxicity of sequential combination therapy of Mitomycin and Bacillus Calmette-Guérin versus Bacillus Calmette-Guérin monotherapy through CTCAE v4.0. Patients have to fill in International Prostate Symptoms Score, NIH-CPSI, PUF questionaries. Every three months patients will be visited and have a cystoscopy. We will hear about self-reported symptoms and we will measure body temperature

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Tubaro, Principal Investigator — Azienda Ospedaliera "Sant'Andrea"

REFERENCES:
- [Background] Solsona E, Madero R, Chantada V, Fernandez JM, Zabala JA, Portillo JA, Alonso JM, Astobieta A, Unda M, Martinez-Pineiro L, Rabadan M, Ojea A, Rodriguez-Molina J, Beardo P, Muntanola P, Gomez M, Montesinos M, Martinez Pineiro JA; Members of Club Urologico Espanol de Tratamiento Oncologico. Sequential combination of mitomycin C plus bacillus Calmette-Guerin (BCG) is more effective but more toxic than BCG alone in patients with non-muscle-invasive bladder cancer in intermediate- and high-risk patients: final outcome of CUETO 93009, a randomized prospective trial. Eur Urol. 2015 Mar;67(3):508-16. doi: 10.1016/j.eururo.2014.09.026. Epub 2014 Oct 6. PMID 25301758
- [Background] Cui J, Wang W, Chen S, Chen P, Yang Y, Guo Y, Zhu Y, Chen F, Shi B. Combination of Intravesical Chemotherapy and Bacillus Calmette-Guerin Versus Bacillus Calmette-Guerin Monotherapy in Intermediate- and High-risk Nonmuscle Invasive Bladder Cancer: A Systematic Review and Meta-analysis. Medicine (Baltimore). 2016 Jan;95(3):e2572. doi: 10.1097/MD.0000000000002572. PMID 26817914
- [Background] Kaasinen E, Wijkstrom H, Rintala E, Mestad O, Jahnson S, Malmstrom PU. Seventeen-year follow-up of the prospective randomized Nordic CIS study: BCG monotherapy versus alternating therapy with mitomycin C and BCG in patients with carcinoma in situ of the urinary bladder. Scand J Urol. 2016 Oct;50(5):360-8. doi: 10.1080/21681805.2016.1210672. Epub 2016 Aug 15. PMID 27603424
- [Derived] Cicione A, Lombardo R, Nacchia A, Franco A, Simone G, Pastore A, Leonardo C, Franco G, Tubaro A, DE Nunzio C. No clinical benefit from sequential combination of mitomycin C plus bacillus Calmette-Guerin (BCG) than BCG alone in the adjuvant treatment of high risk non muscle invasive bladder cancer: result of a planned interim analysis of a prospective randomized trial. Minerva Urol Nephrol. 2024 Aug;76(4):458-466. doi: 10.23736/S2724-6051.24.05777-X. Epub 2024 Jun 5. PMID 38842053